CLINICAL TRIAL: NCT01076686
Title: An Observational Study to Assess the Long-Term Follow-Up of Subjects Who Had Participated in SKY0402 Breast Augmentation Studies
Brief Title: Observational Study to Assess Long-Term Follow-Up of Breast Augmentation Subjects
Status: Completed | Type: Observational
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SKY0402-C-318
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2012-05-14 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2011-12

CONDITIONS: Postoperative Pain
Keywords: Augmentation mammoplasty; Breast augmentation; Postoperative pain; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Bupivacaine and low dose SKY0402
  Interventions: Drug: Questionnaire and Physical Exam
- Bupivacaine and high dose SKY0402
  Interventions: Drug: Questionnaire and Physical Exam
- Bupivacaine
  Interventions: Drug: Questionnaire and Physical Exam
- High dose SKY0402
  Interventions: Drug: Questionnaire and Physical Exam

INTERVENTIONS:
Drug: Questionnaire and Physical Exam — A 10-question survey and a six-item physical exam were completed.

SUMMARY:
A history and physical focused on clinical sequelae of breast implant rupture was completed by patients to assess long-term clinical sequelae of SKY0402 and its relation to the silicon shell.

DETAILED DESCRIPTION:
This was an observational, multicenter study conducted to investigate the long term follow-up of subjects who had been exposed to study drug (either SKY0402, bupivacaine HCl, or both) in prior SKY0402 breast augmentation studies. Specifically, the protocol was designed to elicit any changes in the response of the silicone shell of the implant after exposure to study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participated in either Pacira SKY0402-C-210 or Pacira SIMPLE Breast Augmentation 315 and received a dose of SKY0402, bupivacaine HCl, or both
* Able and willing to comply with all study visits and procedures.
* Able to speak, read, and understand the language of the informed consent, and any other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to study assessments.
* Able and willing to provide written informed consent

Exclusion Criteria:

* Did not receive study drug in either Pacira SKY0402-C-210 or SIMPLE Breast Augmentation 315.
* Has a clinically significant systemic or psychiatric disease that may pose a significant safety risk or diminish a subject's ability to undergo all study procedures and assessments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had been exposed to study drug and had undergone breast augmentation.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

REFERENCES:
- [Derived] Minkowitz HS, Onel E, Patronella CK, Smoot JD. A two-year observational study assessing the safety of DepoFoam bupivacaine after augmentation mammaplasty. Aesthet Surg J. 2012 Feb;32(2):186-93. doi: 10.1177/1090820X11434524. Epub 2012 Jan 11. PMID 22238339

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine and Low Dose SKY0402; Bupivacaine and High Dose SKY0402; Bupivacaine; High Dose SKY0402: Single dose of study drug was injected locally into the breast pockets
Period: Overall Study
Arm/Group | Bupivacaine and Low Dose SKY0402 | Bupivacaine and High Dose SKY0402 | Bupivacaine | High Dose SKY0402
Started | 17 | 14 | 32 | 31
Completed | 17 | 14 | 32 | 31
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine and Low Dose SKY0402 | Bupivacaine and High Dose SKY0402 | Bupivacaine | High Dose SKY0402 | Total
Number analyzed (Participants) | 17 | 14 | 32 | 31 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 32 | 31 | 94
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32 (7.2) | 29 (6.3) | 31 (7.1) | 33 (7.6) | 32 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 32 | 31 | 94
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 14 | 32 | 31 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Breast Implant Rupture
Description: Breast implant rupture and integrity were assessed by reviewing the results of history and physical focused on clinical sequelae of augmentation mammoplasty
Time Frame: 12 to 24 months post surgery
Measure: Number; unit: participants
Arm/Group | Bupivacaine and Low Dose SKY0402 | Bupivacaine and High Dose SKY0402 | Bupivacaine | High Dose SKY0402
Number analyzed (Participants) | 17 | 14 | 32 | 31
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Bupivacaine and Low Dose SKY0402 | Bupivacaine and High Dose SKY0402 | Bupivacaine | High Dose SKY0402
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No